CLINICAL TRIAL: NCT05663190
Title: Localization of Mental Foramen in Relation to Primary Molars A Cone Beam Computed Tomography Study
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Maha Moussa Azab, Lecturer, Fayoum University
Other Study IDs: Mental foramen in children
Record Dates: First submitted 2022-11-23; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Mental Foramen; Cone Beam Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Less than 10-year-old, with cone beam computed tomography imagess with the mental foramen included in field of vision
  Interventions: Other: mental foramen location

INTERVENTIONS:
Other: mental foramen location — location of mental foramen in relation to primary molars

SUMMARY:
. The aim of this study was to determine the location of mental foramen in relation to the lower primary molars using Cone Beam Computed Tomography. And develop simple guidelines for the injection of mental block anaesthesia for children.

DETAILED DESCRIPTION:
Cone Beam Computed Tomographies in a private radiology centre will be screened, Cone Beam Computed Tomography images of less than 10 years old, boys or girls were included in the study. Included Cone Beam Computed Tomography images should have either or both sides of the lower arch in the field of view, with the lower first and second primary molars with no or minimal root resorption. Images with pathologies, fractures, malformations, or abnormal location of teeth that would affect the anatomy or location of mental foramen were excluded from the study.

The vertical diameter of mental foramen was measured on the cross-sectional Cone Beam Computed Tomography images, while the horizontal diameter was measured on the axial scans. The ratio between horizontal and vertical diameters (H:V) was calculated to determine the form of mental foramen

Outcomes

1: vertical and horizontal location of mental foramen in relation to 1ry molars 2. subgroup analysis for the 1st outcome according to age, (< 6 years) vs (> 6 yrs) 3. Mental foramen form according to the Horizontal/Vertical ratio 4. If there is any relation between (location, form, vertical or horizontal dimension of mental foramen) and (Side or Gender)

ELIGIBILITY:
Inclusion Criteria:

Included cone beam computed tomography images should have either or both sides of the lower arch in the field of view, with the lower first and second primary molars with no or minimal root resorption.

Exclusion Criteria:

Images with pathologies, fractures, malformations, or abnormal location of teeth that would affect the anatomy or location of mental foramen were excluded from the study.

Ages: 4 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Cone beam computed tomography lower arch images for less than 10-year-old children
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
horizontal location of mental foramen | Day 1
  the location of mental foramen horizontally in relations to the primary molars (using a a modification of Tebo and Telford classification )
vertical location of mental foramen | Day 1
  the location of mental foramen vertically in relation to the apices of the primary molars (above/at the same level/below) the apices

SECONDARY OUTCOMES:
dimension and form of mental foramen | Day 1
  ratio between horizontal and vertical diameter of the mental foramen

OTHER OUTCOMES:
relation to age | Day 1
  is there is a relation between location of mental foramen and age of a child

CONTACTS AND LOCATIONS:
Overall Officials: maha M azab, Principal Investigator — Fayoum University
Locations (1):
- Alpha Dent, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No